CLINICAL TRIAL: NCT02185014
Title: A Multicenter, Open-Label Study to Evaluate the Long Term Efficacy, Safety, and Tolerability of Repeated Administration of Adalimumab in Subjects With Crohn's Disease
Brief Title: Open Label Study to Evaluate Long Term Efficacy, Safety and Tolerability of Repeated Dosing in Subjects With Crohn's Disease and Who Participated and Successfully Completed M14-115
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-347; 2013-004034-15 (EudraCT Number)
Record Dates: First submitted 2014-07-07; First posted 2014-07-09 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Adalimumab (Other): Participants received open-label adalimumab 40 mg by subcutaneous injection every other week for 40 weeks.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — Adalimumab pre-filled syringe, administered by subcutaneous injection
  Other Names: Humira; ABT-D2E7

SUMMARY:
The purpose of this study is to evaluate the long term efficacy, safety, and tolerability of repeated administration of adalimumab in participants with Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

- Subject successfully enrolled in and completed Study M14-115 (NCT02185014), including the Week 12 ileocolonoscopy.

Exclusion Criteria:

* If the Week 12 (Study M14-115; NCT02185014) colonoscopy shows evidence of dysplasia or malignancy.
* Subject is not in compliance with prior and concomitant medication requirements throughout M14-115 (NCT02185014).
* Subject who developed active Tuberculosis (TB) during M14-115 (NCT02185014), or subject who is non compliant with prophylaxis for latent tuberculosis (TB) initiated per M14-115 (NCT02185014) procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2014-08-12; Primary Completion 2017-11-03 (Actual); Study Completion 2017-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc, Study Director — AbbVie

REFERENCES:
- See also: Related Info — http://rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed Study M14-115 (NCT02185014) were eligible to enroll in this study.
Period: Overall Study
Arm/Group | Adalimumab
Started | 252
Completed | 198
Not Completed | 54
Not completed — Adverse Event | 18
Not completed — Withdrew Consent | 8
Not completed — Lost to Follow-up | 4
Not completed — Lack of Efficacy | 14
Not completed — Requires Alternative/Prohibited Therapy | 5
Not completed — Subject Noncompliance | 1
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Population: Baseline characteristics from lead-in study M14-115 (NCT02185014)
Arm/Group | Adalimumab
Number analyzed (Participants) | 252
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (12.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139
  Male | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 245
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 229
  More than one race | 1
  Unknown or Not Reported | 0
Simplified endoscopic score for crohn's disease (SES-CD) [Mean (Standard Deviation); unit: units on a scale] — The SES-CD evaluates 4 endoscopic variables in 5 segments assessed during ileocolonoscopy. The SES-CD total score is the sum of the 4 endoscopic variable scores and range from 0 to 56, where higher scores indicate more severe disease.
  units on a scale | 14.2 (6.74)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Endoscopic Improvement at Week 40 in Participants With Endoscopic Improvement at Week 0
Description: Endoscopic improvement defined as a simple endoscopic score for Crohn's Disease (SES-CD) score of ≤4 and at least a 2-point reduction compared with Study M14-115 (NCT02185014) Baseline and no subscore greater than 1 in any individual endoscopic variable. The SES-CD evaluates 4 endoscopic variables (ulcer size ranging from 0 [none] to 3 [very large]; ulcerated surface ranging from 0 [none] to 3 [>30%]; affected surface ranging from 0 [none] to 3 [>75%], and narrowing ranging from 0 [none] to 3 [cannot be passed]) in 5 segments assessed during ileocolonoscopy (ileum, right colon, transverse colon, sigmoid and left colon, and rectum). The Total Score is the sum of the 4 endoscopic variable scores and range from 0 to 56, where higher scores indicate more severe disease. Nonresponder imputation (NRI) was used for missing data.
Time Frame: Week 40
Population: All enrolled participants who had endoscopic improvement at Week 0 in Study M14-347 (end of lead-in Study M14-115 [NCT02185014])
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 76
percentage of participants | 31.6 [21.1 to 42.0]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until 70 days after the last dose of study drug (up to 48 weeks).
Arm/Group | Adalimumab
All-Cause Mortality (participants affected / at risk) | 0/252
Serious Adverse Events (participants affected / at risk) | 27/252
Other Adverse Events (participants affected / at risk) | 63/252
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adalimumab (N=252)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1)
CROHN'S DISEASE (Gastrointestinal disorders) | 14 (16)
ILEAL STENOSIS (Gastrointestinal disorders) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 3 (3)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 4 (4)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1)
ANAL ABSCESS (Infections and infestations) | 3 (3)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adalimumab (N=252)
CROHN'S DISEASE (Gastrointestinal disorders) | 30 (31)
NAUSEA (Gastrointestinal disorders) | 15 (21)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 13 (13)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 18 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2014-12-04): https://cdn.clinicaltrials.gov/large-docs/14/NCT02185014/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/14/NCT02185014/SAP_001.pdf